CLINICAL TRIAL: NCT02397317
Title: Stereotactic Prostate Adaptive Radiotherapy Utilising Kilovoltage Intrafraction
Brief Title: Stereotactic Prostate Adaptive Radiotherapy Utilising Kilovoltage Intrafraction Monitoring
Acronym: SPARK
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sydney (Other)
Collaborators: Trans Tasman Radiation Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TROG 15.01 SPARK; TROG 15.01 (Other: Trans Tasman Radiation Oncology Group)
Record Dates: First submitted 2015-03-09; First posted 2015-03-24 (Estimated); Last update posted 2017-06-22 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Multi-fraction SABR (Experimental): All participants will receive Multi-Fraction SABR; 36.25 Gy (PTV D95) in 5 Fractions within 2-5 weeks
  Interventions: Radiation: Multi-fraction SABR

INTERVENTIONS:
Radiation: Multi-fraction SABR — All participants will receive Multi-Fraction SABR; 36.25 Gy (PTV D95) in 5 Fractions within 2-5 weeks

SUMMARY:
The SPARK trial is testing the use of Kilovoltage Intrafraction Monitoring in prostate cancer patients being treated with Stereotactic Prostate Adaptive Radiotherapy. The researchers expect this trial to result in better targeted prostate cancer patient outcomes with lower toxicity. The potential application of Kilovoltage Intrafraction Monitoring to other tumour sites will pave the way for additional trials with Australasian radiation oncology leading the world.

DETAILED DESCRIPTION:
Most linear accelerators used to treat cancer patients today are equipped with fixed X-ray imagers which are typically used to take images of a tumour before a patient receives radiotherapy. A new technology, known as Kilovoltage Intrafraction Monitoring has recently emerged which allows images of a tumour to be taken in real-time while the treatment is occurring. The advantage of Kilovoltage Intrafraction Monitoring is that it enables strategies such as patient shifting or beam shifting during treatment which could potentially improve the accuracy of the treatment and reduce the patient's side effects. In addition, due to the accuracy of Kilovoltage Intrafraction Monitoring in targeting tumours, the number of treatment sessions this group of patients will require will be reduced to five as opposed to the 40 sessions required using more conventional treatment methods.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven prostate adenocarcinoma
2. Low or intermediate risk disease as defined by:

   * Low Risk: All of PSA<10 ng/mL, Gleason Grade 6 AND Stage T1 or T2a
   * Intermediate Risk: Any or all of PSA 10-20 ng/mL, Gleason Grade 7 OR Stage T2b-c
   * Absence of high risk features (PSA>20, T3-4, N1 or M1 disease, Gleason score 8-10) (PSA must be within 3 months prior to enrolment)
3. ECOG Performance status 0-2
4. Suitable for definitive external beam radiotherapy (IMRT or VMAT)
5. Ability to have three gold fiducial markers placed in the prostate
6. Six month course of androgen deprivation therapy allowed at clinician discretion.
7. Available for follow up for a minimum of 2 years (up to 3 years)

Exclusion Criteria:

1. Lymph node irradiation
2. Any other systemic anti-prostate cancer therapy (i.e. non-ADT) both proven in the metastatic setting and investigational (e.g. docetaxel, enzalutamide)
3. Artificial hip(s) (Unable to visualise markers through prosthesis)
4. Prostate volume > 90 cm3 measured from the CT scan
5. Patient lateral dimension >40cm as measured at the level of the prostate from the CT scan
6. Suboptimal fiducial markers placement for treatment utilising KIM as assessed by a medical physicist by measuring marker positions from the CT scan
7. Fiducial migration or fewer than 3 fiducials present in the CT scan

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Accumulated patient dose distributions will be determined via paired controls by comparing the measured treatment accuracy and dose with KIM and those that would have been delivered in the absence of KIM | up to 36 months

SECONDARY OUTCOMES:
Patient treatment outcomes determined by assessing Biochemical-clinical failure (BCF) | up to a maximum of 36 months.
Patient treatment outcomes determined by assessing acute and late toxicity grade 3 or higher (using CTCAE version 4) | Weekly during treatment, then two weeks, six weeks and 6 months post treatment
Patient treatment outcomes determined by assessing patient-reported outcomes | 12 and 24 months after treatment
The patient's perception of KIM will be quantified using an adapted SAT-RAR survey, an instrument that has previously been used to assess patient perceptions on technological innovations in radiotherapy and respiratory gating. | up to 36 months
Targeting accuracy through measuring the final geometric accuracy with and without the KIM gating procedure | up to 36 months
Radiation therapists feedback on KIM will be quantified using a survey which will obtain specific information about the impact of the KIM system and SPARK on education, patient workflow, clinical impact and user confidence | up to 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul Keall, Study Chair — University of Sydney; Jarad Martin, Study Chair — Calvary Mater Newcastle
Locations (5):
- Australia (5):
  - Calvary Mater Newcastle, Newcastle, New South Wales
  - Liverpool Cancer Therapy Centre, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - The Crown Princess Mary Cancer Centre Westmead, Sydney, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chrystall D, Mylonas A, Hewson E, Martin J, Keall P, Booth J, Nguyen DT. Deep learning enables MV-based real-time image guided radiation therapy for prostate cancer patients. Phys Med Biol. 2023 Apr 26;68(9). doi: 10.1088/1361-6560/acc77c. PMID 36963116
- [Derived] Hewson EA, Nguyen DT, O'Brien R, Poulsen PR, Booth JT, Greer P, Eade T, Kneebone A, Hruby G, Moodie T, Hayden AJ, Turner SL, Hardcastle N, Siva S, Tai KH, Martin J, Keall PJ. Is multileaf collimator tracking or gating a better intrafraction motion adaptation strategy? An analysis of the TROG 15.01 stereotactic prostate ablative radiotherapy with KIM (SPARK) trial. Radiother Oncol. 2020 Oct;151:234-241. doi: 10.1016/j.radonc.2020.08.010. Epub 2020 Aug 20. PMID 32828839
- [Derived] Keall P, Nguyen DT, O'Brien R, Booth J, Greer P, Poulsen P, Gebski V, Kneebone A, Martin J. Stereotactic prostate adaptive radiotherapy utilising kilovoltage intrafraction monitoring: the TROG 15.01 SPARK trial. BMC Cancer. 2017 Mar 8;17(1):180. doi: 10.1186/s12885-017-3164-1. PMID 28270121